CLINICAL TRIAL: NCT03454503
Title: Evaluation of Generic Imatinib in a Real-World Setting Among Chronic Myeloid Leukemia Patients in Egypt
Brief Title: Effectiveness and Safety Study of Generic Imatinib in Chronic Myeloid Leukemia Patients in Egypt
Status: Completed | Type: Observational
Sponsor: Hikma Pharmaceuticals LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: CRC-EGY-2016-05
Record Dates: First submitted 2018-02-26; First posted 2018-03-06 (Actual); Last update posted 2021-02-23 (Actual); Status verified 2020-03

CONDITIONS: Philadelphia Chromosome-positive Chronic Myeloid Leukemia in Chronic Phase
Keywords: Imatinib; Generic Imatinib; Leukemia; Chronic myeloid leukemia; Philadelphia chromosome-positive; Chronic phase; Observational study; Switched patients; Tyrosine kinase inhibitor
MeSH Terms: conditions — Leukemia; Leukemia, Myelogenous, Chronic, BCR-ABL Positive | interventions — Imatinib Mesylate

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- First cohort: Newly diagnosed patients
  Interventions: Drug: Imatinib
- Second cohort: Patients switched from reference product (Glivec® )
  Interventions: Drug: Imatinib

INTERVENTIONS:
Drug: Imatinib — Film coated tablet contains 400 mg imatinib (as mesilate)
  Other Names: Carcemia®

SUMMARY:
The purpose of this observational study is to evaluate the effectiveness and safety of generic imatinib under usual clinical practice in patients of Philadelphia chromosome-positive (Ph+) chronic myeloid leukemia (CML) patients in chronic phase (CP) in Egypt

DETAILED DESCRIPTION:
An observational, multi-center, prospective cohort study to assess the effectiveness and safety of generic Imatinib (Carcemia®) in patients with Ph+ CML who are newly diagnosed or patients who will be switched from the reference product (Glivec® ) to Carcemia® where treatment will be prescribed by the investigator in accordance with clinical practice where no visits or intervention(s) additional to the daily practice will be performed.

Eligible Ph+ CML patients in both cohorts will be followed up for a total of 18 months.

ELIGIBILITY:
Inclusion Criteria:

First cohort (newly diagnosed patients):

* Age ≥18 years
* Newly diagnosed patients with Ph+ CML in CP, with or without the presence of other cytogenetic abnormalities at the time of diagnosis
* Treatment naïve patients with confirmed diagnosis within 3 months of study enrolment
* Levels of liver aminotransferases and serum bilirubin ≤ 2 times the upper limit of the normal range, and serum creatinine ≤1.5 times the upper limit of the normal range
* Written informed consent

Second cohort (switched patients):

* Age ≥18 years
* Ph+ CML patients in CP currently treated with Glivec®, with or without the presence of other cytogenetic abnormalities at the time of switch
* Levels of liver aminotransferases and serum bilirubin ≤ 2 times the upper limit of the normal range and serum creatinine ≤1.5 times the upper limit of the normal range
* Written informed consent

Exclusion Criteria:

* CML in accelerated phase (AP) at enrollment except patients in AP with the presence of other cytogenetic abnormalities at the time of diagnosis
* CML in BP at enrollment
* Patients who meet any of the contraindications to the administration of the study drug according to the approved Summary of Product Characteristics

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be recruited from 2 sites in Egypt
Sampling Method: Non-Probability Sample
Enrollment: 173 (Actual)
Dates: Start 2018-05-13 (Actual); Primary Completion 2020-12-28 (Actual); Study Completion 2020-12-28 (Actual)

PRIMARY OUTCOMES:
Proportion of patients who achieve and maintain major molecular response (MMR) | 12 months
  Major molecular response (MMR) is measured using real-time quantitative polymerase chain reaction (RQ-PCR) test and is defined as BCR-ABL1 ≤ 0.1%

SECONDARY OUTCOMES:
Incidence of adverse events (AEs) and serious adverse events (SAEs) to generic Imatinib (Carcemia®) | 18 months
  Number, type, severity and frequency of adverse events (AEs), serious AEs (SAEs), and clinically relevant changes in laboratory tests according to laboratory reference ranges
Progression free survival (PFS) | 18 months
  Proportion of CML patients who will not experience disease progression from enrollment to 18 months study endpoint.
Event free survival (EFS) | 18 months
  Proportion of CML patients who will not experience event from enrollment to 18 months study endpoint
Survival without blastic phase (BP) | 18 months
  Proportion of CML patients who will not experience blastic phase (BP) from enrollment to 18 months study endpoint.
Overall survival (OS) | 18 months
  Proportion of CML patients who will not die till 18 months study endpoint.
Complete cytogenetic response (CCgR) | 12 months
  Proportion of CML patients who will achieve no Ph+ metaphases at 12 months study endpoint by conventional cytogenetics and/or FISH test.
Complete molecular response (CMR) | 12 months
  Proportion of CML patients who will achieve undetectable BCR-ABL mRNA transcripts by RQ-PCR test in two consecutive blood samples of adequate quality.
Health-Related Quality of Life (HRQoL) | 18 months
  Mean change in Health-Related Quality of Life (HRQoL) utilizing EORTC QOLCML24 questionnaire throughout treatment visits
Treatment compliance on generic Imatinib | 18 months
  Evaluated by identifying the frequency of not taking the medications as prescribed and the reasons. The decision on non-compliance is based on the treating physician's judgment.

CONTACTS AND LOCATIONS:
Locations (1):
- National Cancer Institute (NCI), Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No